CLINICAL TRIAL: NCT05593302
Title: The Effectiveness of Trauma Focused Art Therapy: a Multiple Baseline Single Case Experimental Design
Brief Title: The Effectiveness of Trauma Focused Art Therapy
Acronym: TFAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HAN University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Suzanne Haeyen, dr. Suzanne Haeyen, HAN University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TFAT SU1424 -101
Record Dates: First submitted 2022-10-12; First posted 2022-10-25 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-06

CONDITIONS: Trauma; Psychological; Art Therapy
Keywords: Art Therapy; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Multiple baseline single case experimental design (MBSCED) wherein all patients are first assigned to the control condition (or control period) and are then assigned to the intervention condition (or intervention period) and finally the follow-up period (control period). Patients are randomized for the time (t) at which they start with the intervention. The Single-Case Reporting Guideline In BEhavioural Interventions (SCRIBE) recognizes the MBSCED as an experimental design (doi: 10.1016/j.jclinepi.2016.04.006).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Control Period - Intervention Period (Experimental): Multiple baseline single case experimental design wherein all patients are first assigned to the control condition (or control period) are then assigned to the intervention condition (or intervention period) and finally to the follow-up period (control period). Patients are randomized for the time (t) at which they start with the intervention.
  Interventions: Behavioral: Trauma-Focused Art Therapy (TFAT)

INTERVENTIONS:
Behavioral: Trauma-Focused Art Therapy (TFAT) — Individual Trauma Focused Art Therapy (TFAT) consisting of 10 sessions. Each session lasts 60 minutes. Sessions are aimed at trauma recovery using visual art therapy. The sessions cover an introduction, making pieces of artwork, and reflection. Three phases can be distinguished:
  Phase 1: 'stabilization and symptom reduction', i.e. exploring traumatic and positive memories, imagining a lifecourse, and expressing a safe haven (4 sessions).
  Phase 2:'uttering and expressing memories', i.e. expressing chosen memories by making 5 pieces of artwork. Materials that can be used include clay, paint, graphite pencil or crayons and if needed with support of imagination using relevant photographs or objects (5 sessions).
  Phase 3: 'integration and meaning attribution', i.e. ordering and assembling of the 5 pieces of artwork. Patients are asked to appraise the memories in the here-and-now present (c.f. mindfulness-based cognitive therapy) (1 session).

SUMMARY:
More than 30% of patients with trauma-related complaints do not benefit from prescribed treatments. This concerns patients who have either a poor verbal memory or who are unable or do not wish to talk about their experiences.

In clinical practice, trauma-oriented art therapy appears to be an appropriate treatment. The visual, tangible, experiential character of art therapy is in line with the often wordless, visual and sensory nature of trauma.

Art therapy aims to contribute to achieving personal goals through the use of visual materials and techniques. This approach has been insufficiently examined. Treatment of refugees with Trauma-Focused Art Therapy has previously been shown to be feasible in clinical practice and acceptable to patients.

Using a Mixed Method design, the researchers aim to measure the effect of this protocol in specialized mental health care and the experience of patients with regard to their personal recovery.

DETAILED DESCRIPTION:
INTRODUCTION:

About four in five people experience one or more distressing events in their lives. Ten percent of people subsequently develop post-traumatic stress disorder (PTSD). About 1.3 million people in the Netherlands will therefore have to deal with the consequences of PTSD at some point. PTSD is an anxiety disorder and causes serious complaints of re-experience, avoidance and increased irritability as a result of exposure to one or more traumatic events. The disorder causes significant distress or impairment in social, occupational, or other important areas of functioning,

According to the Anxiety Disorders Guideline and the guidelines of the National Institute for Health and Care Excellence (NICE), Cognitive Behavioral Therapy (CBT) and Eye Movement Desensitization and Reprocessing (EMDR) are the preferred treatments for PTSD. However, these interventions do not work for everyone - more than a third of patients do not benefit. This includes patients with very severe traumatization, with poor verbal memory and patients who are unable or patients who find it difficult to talk about the traumatic experiences.

Practice shows that art therapy (AT) offers an appropriate treatment for these patients. This is because the visual, tactile and experiential nature of AT fits well with the often wordless, visual and sensory nature of traumatic memories. Trauma-focused AT provides access to memories and emotions, can help to put these into words, and can be a possible preliminary stage (pretherapy) for other trauma-focused treatments (such as EMDR, CBT or NET).

Patient representatives underline the availability of trauma treatment based on AT because they believe that it offers an essential alternative to the usual verbal, often cognitive therapeutic approach. In addition, the Improvement Report Posttraumatic Stress Disorders from the Netherlands Healthcare Institute mentions, as one of the most important points for improvement, that more people with PTSD should receive specific trauma-oriented treatment.

AT is one of the arts therapies: The treatment tradition of arts therapies spans about a century and includes the disciplines: visual, drama, dance, music and psychomotor therapy. AT works through the use of numerous visual materials, methods and techniques to give meaning to past events and to gain more control over one's own life.

AT distinguishes itself from other treatments by its experiential approach and by the visible and tangible nature of the process and product of the treatment. Acting, doing and experiencing with visual material removes the feeling of powerlessness, increases the sense of control and the sense of self-worth. Working with visual material triggers emotions: it allows access to traumatic memories and emotions (AT makes it possible to express and shape, integrate and accommodate traumatic memories in a safe and staged way. The result of the visual work is visible, tangible and has a lasting character. This allows one to literally distance themselves from the emotion, integrate it cognitively and assign meaning. AT is more often applied in practice with good results according to patients and professionals, but has been insufficiently examined.

A Trauma-Focused Art Therapy protocol was previously developed. In a pilot study with patients with early childhood traumatization, this protocol was found to be acceptable, feasible and applicable. This protocol lends itself to transferring this method between art therapists, but has not yet been further investigated for effectiveness. In this project, this protocol is implemented, tested and evaluated by patients and professionals.

The Trauma-Focused Art Therapy protocol offers opportunities to improve accessibility, quality and effectiveness of trauma treatment, because patients who would otherwise not be treated or who would receive long-term treatments without results, now receive appropriate treatment. This concerns a short-term, individual trauma-focused AT consisting of 10 sessions (60 min.) in three phases (I: Stabilization and symptom reduction; II: Trauma processing; III: integration and attribution of meaning). After the first phase of getting acquainted, creating safety and determining a list of memories, phase 2 works on expressing and shaping positive and negative feelings, memories and thoughts. Phase 3 focuses on reordering, merging and finalizing the AT.

RESEARCH QUESTIONS:

Is the Trauma-Focused Art Therapy protocol an effective treatment of patients' trauma-related complaints

How do patients and art therapists experience this method?

OBJECTIVES:

The aim of this research is to gain insight into the effectiveness and functioning of trauma-focused AT. This contributes to evidence about the effectiveness of trauma treatment.

The aim is to better align trauma treatment with patients' needs to work on personal recovery in a different way. The protocol is tested in practice with the help of patients and professionals on: symptom reduction and psychological health.

HYPOTHESIS:

Art therapy offers an appropriate treatment for the group of multiple and long-term traumatized patients, who avoid and/or have difficulty talking about traumatic memories, because the visual and tangible character of art therapy seems to match the often wordless, visual and sensory nature of traumatic memories.Trauma-focused art therapy reduces PTSD symptoms (avoidance, arousal and re-experiencing) and depression (if there is comorbidity) and enhances self-confidence/self-esteem, mental resilience and positive health.

ELIGIBILITY:
Inclusion Criteria:

* Having trauma-related symptoms ((i.e. nightmares, flashbacks, persistent fatigue or depression, anxiety in regards to specific triggers, sleep disorders)
* Being eligible for art therapy on discretion of multidisciplinary treatment panel (consisting of, for example. a psychiatrist, psychologists, sociotherapists, and art therapists)
* Being motivated to work on traumatic memories

Exclusion Criteria:

* Psychosis or acute crisis
* intellectual disability (precluding the filling out of questionnaires).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Self-expression and Emotion Regulation in Art Therapy Scale | 16-18 repeated measures of emotional self-expression and regulation, i.e. weekly over the course of 18 weeks (3-5 weeks control period + 10 weeks intervention + 3 weeks follow-up))
  Self-expression and Emotion Regulation in Art Therapy Scale (SERATS): Assessment of emotional self-expression and regulation during therapy with 9 5-point scale items

SECONDARY OUTCOMES:
Rosenberg Self-Esteem Scale | 16-18 repeated measures of self-esteem, i.e. weekly over the course of 18 weeks (3-5 weeks control period + 10 weeks intervention + 3 weeks follow-up))
  Rosenberg Self-Esteem Scale (RSES): Self-esteem assessed with ten 4-point scale items
Resilience Scale | 16-18 repeated measures of mental resiliency, i.e. weekly over the course of 18 weeks (3-5 weeks control period + 10 weeks intervention + 3 weeks follow-up))
  Resilience Scale (RS): Mental resiliency i.e. how patients cope with challenges, drawbacks, and distressing circumstances assessed with 25 4-point scale items
Beck Depression Inventory | 16-18 repeated measures of depression severity, i.e. weekly over the course of 18 weeks (3-5 weeks control period + 10 weeks intervention + 3 weeks follow-up))
  Beck Depression Inventory (BDI): Severity of depression scored in the domains of affective, cognitive and somatic symptoms assessed with 21 4-point scale items
Mental Health Continuum Short Form (MHC-SF) | 16-18 repeated measures of positive mental health, i.e. weekly over the course of 18 weeks (3-5 weeks control period + 10 weeks intervention + 3 weeks follow-up))
  Mental Health Continuum Short Form (MHC-SF): positive mental health in the domains of emotional, psychological, and social wellbeing using 14 items
Post-traumatic stress disorder Check List | Change from baseline PTSD symptoms at 15 weeks (after completion of intervention)
  Post-traumatic stress disorder Check List (PCL): screener of symptoms of PTSD using 20 items based on the Diagnostic and Statistical Manual 5th edition (DSM-5)

CONTACTS AND LOCATIONS:
Overall Officials: Christine De Vries, Msc., Study Director — HAN University of Applied Sciences
Locations (1):
- HAN University of Applied Sciences, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We will not make IPD directly available, but rather indirectly through a description of the meta-data and contact information of the principal investigator, to whom data requests can be sent.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the main paper until 10 years after this publication.
Access Criteria: The principal investigator will investigate whether requests are reasonable and feasible and adhere to ethical considerations.

REFERENCES:
- [Derived] Heijman J, Wouters H, Schouten KA, Haeyen S. Effectiveness of trauma-focused art therapy (TFAT) for psychological trauma: study protocol of a multiple-baseline single-case experimental design. BMJ Open. 2024 Jan 29;14(1):e081917. doi: 10.1136/bmjopen-2023-081917. PMID 38286685